CLINICAL TRIAL: NCT05336253
Title: The EVERYbody Project-Connect: A Randomized-Controlled Study Comparing Active and Passive Inclusive Online Body Image Content for College Students
Brief Title: Online Expert Peer Facilitation of the EVERYbody Project
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Western Washington University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Prevention
Other Study IDs: 4482EX21
Record Dates: First submitted 2022-03-01; First posted 2022-04-20 (Actual); Last update posted 2023-12-18 (Actual); Status verified 2023-12

CONDITIONS: Body Image; Eating Disorder Symptom; Weight Bias
Keywords: Dissonance Intervention; Body Image; Eating Disorders Prevention
MeSH Terms: conditions — Weight Prejudice

STUDY DESIGN:
Intervention Model Description: Participants will be randomized on a 1:1 basis through survey software to the EVERYbody Project-Connect or the self-help workbook condition
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- EVERYbody Project-Connect Online Program (Experimental): Three weekly 90-minute online group sessions facilitated by expert peer leaders. Retains key dissonance activities and the inclusivity focus of the original EVERYbody Project (e.g., expanded gender focus, critically discussing the impact of limited diversity representation in cultural appearance norms). Additional activities were added, including an increased focus on body compassion (self-acceptance) and weight neutrality content to target weight bias.
  College students with body image interest and lived or academic diversity and advocacy experience will complete 16 hours of training to become expert peer leaders. Training includes observation, practice, and feedback on using the program manual and managing groups. Students will self-assess and be evaluated by the primary trainer on facilitation readiness. Only peer leaders with sufficient expertise will be invited to facilitate groups.
  Interventions: Behavioral: EVERYbody Project-Connect
- Self-Help Workbook (Active Comparator): In this time-matched comparison intervention, participants will be provided with an online copy of The Body Is Not An Apology Workbook by author and activist Sonya Renee Taylor (2021). Weekly emails will assign workbook activities to complete on their own (90 minutes per week for three weeks). This low-dissonance comparison intervention covers many of the same topics within the EVERYbody Project-Connect (body acceptance and scrutinizing the diversity within body ideals) and its activities include reflective writing and drawing exercises to challenge media messages around bodies, identify systems of oppression underpinning body messages, challenge body stereotypes, and make peace with your own body. Activities within the workbook are considered low-dissonance since they will be done privately and not shared.
  Interventions: Behavioral: Self-Help Workbook

INTERVENTIONS:
Behavioral: EVERYbody Project-Connect — 3-week dissonance-based, group, online body image program (4.5 hours total)
  Arms: EVERYbody Project-Connect Online Program
Behavioral: Self-Help Workbook — Time-matched 3-week passive, individual workbook condition (4.5 hours total)
  Arms: Self-Help Workbook

SUMMARY:
This randomized-controlled trial examines an online dissonance-based body image program for college students called the EVERYbody Project-Connect. The online (videoconferencing) intervention will be delivered using expert peer leaders in three 90-minute weekly sessions. Expert peer leaders for the EVERYbody Project-Connect are college students with lived and/or academic expertise within both body image and diversity and equity domains who are trained and screened for facilitation readiness. The comparison intervention is a passive, time-matched self-help condition using The Body Is Not An Apology Workbook by Sonya Renee Taylor. Both interventions explore diversity and representation within sociocultural body image pressures and provide tools for body acceptance.

The study is open to all college students in a universal prevention and risk factor reduction framework. Outcomes will be assessed before and after the three weeks of intervention and at three-month follow-up.

DETAILED DESCRIPTION:
To date, three completed trials of the EVERYbody Project demonstrate that a gender-inclusive, diversity-focused, dissonance based group program can improve eating disorder risk factors and body image among college students. Through active written and verbal exercises and discussion, students directly challenge the cultural messages that appearance should fit within a narrow set of "ideals," critiquing the diversity representation within appearance ideals and incorporating new strategies for body acceptance.

Although peer (aka student to student) facilitation is commonly used for delivering dissonance-based body image interventions, an open training model (where all interested students are eligible to facilitate after training) may not be the most beneficial for leading inclusivity-focused body image groups. Research suggests that the EVERYbody Project is most effective when delivered by either (1) professional facilitators (faculty or staff with body image expertise), or (2) expert peer leaders (college students with lived or academic expertise in both body image and diversity topics who are screened for facilitation readiness during training).

The current trial explores an online adaptation of this program. The EVERYbody Project-Connect was created from the original program after end-user piloting with college students. The resulting program consists of three 90-minute weekly sessions delivered by expert peer leaders over a secure videoconferencing platform. Expert peer facilitators will complete a 16-hour online training and be screened for facilitation readiness before being approved to lead the intervention. Participants will be randomized on a 1:1 basis to receive the EVERYbody Project-Connect or a time-matched, low-dissonance self-help workbook intervention. Participants in this comparison intervention will be provided with an online copy of The Body Is Not An Apology Workbook by author and activist Sonya Renee Taylor and given weekly assignment instructions (90 minutes of activities each week for three weeks). Workbook activities will be completed on their own as a passive self-help intervention.

College students in the Pacific Northwest United States will be invited to participate in this study (universal intervention target, gender inclusive). Outcome assessment includes a comparison of changes in eating disorder risk factors, eating disorder symptoms, and related constructs across conditions over time (from pre- to post-intervention and through 3-month follow-up). Program satisfaction will be assessed at post-intervention, and program application will be evaluated both post-intervention and at follow-up.

ELIGIBILITY:
Inclusion Criteria:

* Current college students (enrolled with university email address)

Exclusion Criteria:

* None

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 170 (Actual)
Dates: Start 2022-01-14 (Actual); Primary Completion 2023-08-30 (Actual); Study Completion 2023-08-30 (Actual)

PRIMARY OUTCOMES:
Internalized appearance norms | Change from baseline through post-intervention (3 weeks later) and follow-up (3 months)
  Internalization subscales from the Sociocultural Attitudes Toward Appearance Questionnaire-4 (SATAQ-4). Average of 10 items; higher scores indicate greater internalization of cultural messages surrounding appearance and attractiveness.
Body dissatisfaction | Change from baseline through post-intervention (3 weeks later) and follow-up (3 months)
  Satisfaction and Dissatisfaction with Body Parts Scale (SDBPS). Average of 9 items; higher scores equal greater dissatisfaction with nine body parts that are commonly endorsed as concerning (e.g., stomach, thighs, hips). The scale will be reverse scored from the original.
Eating disorder pathology | Change from baseline through post-intervention (3 weeks later) and follow-up (3 months)
  8-item version of the Eating Disorders Examination Questionnaire (EDE-Q8). Average of 8 items for Global Score; higher scores equal greater frequency and severity of disordered attitudes and behaviors over the past month.
Negative affect | Change from baseline through post-intervention (3 weeks later) and follow-up (3 months)
  Fear, guilt, and sadness subscales of the Positive and Negative Affect Schedule-Revised (PANAS). Average of 20 items; higher scores equal greater negative emotion.

SECONDARY OUTCOMES:
Weight bias | Change from baseline through post-intervention (3 weeks later) and follow-up (3 months)
  Anti-fat attitudes scale (AFAS). Average of 5 items; higher scores equal greater negative stereotypes about fat people and fear of fat.
Positive body image | Change from baseline through post-intervention (3 weeks later) and follow-up (3 months)
  Body Appreciation Scale-2 (BAS-2). Average of 10 items; higher scores equal greater body positivity.

OTHER OUTCOMES:
Week 1 weight bias change | Assessed at Week 1 of intervention (one week after baseline)
  Interim assessment of weight bias after Week 1 of the 3-week interventions using the Anti-fat attitudes scale (AFAS). Change from baseline to Week 1 will be used to predict post-intervention and follow-up outcomes.
Week 1 internalization change | Assessed at Week 1 of intervention (one week after baseline)
  Interim assessment of internalization of appearance norms after Week 1 of the 3-week interventions using the Sociocultural Attitudes Toward Appearance Questionnaire-4 (SATAQ-4). Change from baseline to Week 1 will be used to predict post-intervention and follow-up outcomes.
Program satisfaction | Assessed at post-intervention (three weeks after baseline)
  Four Likert scale items about enjoyment (e.g., "I enjoyed the EVERYbody Project") averaged for total satisfaction score (higher score equals greater satisfaction). Three open-ended questions (e.g., "Was any part of the EVERYbody Project particularly helpful/useful? If so, which part and why?") coded for themes.
Program application | Assessed at post-intervention (three weeks after baseline) and follow-up (3 months)
  Three Likert questions to gauge the application of new information (e.g., "How often do you think about the things you learned in the EVERYbody Project?"). Items will be averaged for a total application score (higher scores equaling more frequent application). One open-ended question on the 3-month follow-up survey only to report any other ways the EVERYbody Project has impacted the participant recently.

CONTACTS AND LOCATIONS:
Locations (1):
- Western Washington University, Bellingham, Washington, United States

IPD SHARING:
Plan to Share IPD: Yes
Data and other materials will be made available following reasonable request to study Principal Investigator. All outcome data will be included in data sharing. Socio-demographic characteristics will be collapsed into broader categories to protect participant identity.
  Other study materials, including intervention manuals, will be housed on the Principal Investigator's Open Science Framework page, where URLs will be made publicly available.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Data will be made available three months after data collection is complete.
URL: http://osf.io/x3k7v/?view_only=c9dbd31a4ad94a08b16421d719bc0fac

REFERENCES:
- [Background] Ciao AC, Munson BR, Pringle KD, Roberts SR, Lalgee IA, Lawley KA, Brewster J. Inclusive dissonance-based body image interventions for college students: Two randomized-controlled trials of the EVERYbody Project. J Consult Clin Psychol. 2021 Apr;89(4):301-315. doi: 10.1037/ccp0000636. PMID 34014692
- [Background] Ciao AC, Ohls OC, Pringle KD. Should body image programs be inclusive? A focus group study of college students. Int J Eat Disord. 2018 Jan;51(1):82-86. doi: 10.1002/eat.22794. Epub 2017 Nov 6. PMID 29105805
- [Background] Schaefer LM, Burke NL, Thompson JK, Dedrick RF, Heinberg LJ, Calogero RM, Bardone-Cone AM, Higgins MK, Frederick DA, Kelly M, Anderson DA, Schaumberg K, Nerini A, Stefanile C, Dittmar H, Clark E, Adams Z, Macwana S, Klump KL, Vercellone AC, Paxton SJ, Swami V. Development and validation of the Sociocultural Attitudes Towards Appearance Questionnaire-4 (SATAQ-4). Psychol Assess. 2015 Mar;27(1):54-67. doi: 10.1037/a0037917. Epub 2014 Oct 6. PMID 25285718
- [Background] Stice E, Shaw H, Burton E, Wade E. Dissonance and healthy weight eating disorder prevention programs: a randomized efficacy trial. J Consult Clin Psychol. 2006 Apr;74(2):263-75. doi: 10.1037/0022-006X.74.2.263. PMID 16649871
- [Background] Berscheid, E., Hatfield [Walster], E., & Bohrnstedt, G. (1973). The happy American body: A survey report. Psychology Today, 7, 119-131.
- [Background] Watson, D., & Clark, L. A. (1992). Affects separable and inseparable: On the hierarchical arrangement of the negative affects. Journal of Personality and Social Psychology, 62, 489-505. http://dx.doi.org/10.1037/ 0022-3514.62.3.489
- [Background] Kliem S, Mossle T, Zenger M, Strauss B, Brahler E, Hilbert A. The eating disorder examination-questionnaire 8: A brief measure of eating disorder psychopathology (EDE-Q8). Int J Eat Disord. 2016 Jun;49(6):613-6. doi: 10.1002/eat.22487. Epub 2015 Dec 29. PMID 26711183
- [Background] Becker CB, Stice E. From efficacy to effectiveness to broad implementation: Evolution of the Body Project. J Consult Clin Psychol. 2017 Aug;85(8):767-782. doi: 10.1037/ccp0000204. PMID 28726480
- [Background] Ciao AC, Latner JD, Brown KE, Ebneter DS, Becker CB. Effectiveness of a peer-delivered dissonance-based program in reducing eating disorder risk factors in high school girls. Int J Eat Disord. 2015 Sep;48(6):779-84. doi: 10.1002/eat.22418. Epub 2015 May 8. PMID 25959408
- [Background] Crandall, C., & Biernat, M. (1990). The Ideology of Anti-Fat Attitudes. Journal of Applied Social Psychology, 20(3), 227-243.
- [Background] Faul F, Erdfelder E, Lang AG, Buchner A. G*Power 3: a flexible statistical power analysis program for the social, behavioral, and biomedical sciences. Behav Res Methods. 2007 May;39(2):175-91. doi: 10.3758/bf03193146. PMID 17695343
- [Background] Tylka TL, Wood-Barcalow NL. The Body Appreciation Scale-2: item refinement and psychometric evaluation. Body Image. 2015 Jan;12:53-67. doi: 10.1016/j.bodyim.2014.09.006. Epub 2014 Oct 21. PMID 25462882
- [Background] Taylor, S. R. (2021). The Body Is Not An Apology Workbook: Tools for Living Radical Self-Love. Beret-Koehler Publishers, Inc.